CLINICAL TRIAL: NCT02256917
Title: Prospective, Open-label, Multi-centre Phase 3b Study to Assess the Efficacy and Safety of Personalized Prophylaxis With Human-cl rhFVIII in Previously Treated Adult Patients With Severe Haemophilia A
Brief Title: Assess the Efficacy and Safety of Personalized Prophylaxis Human-cl rhFVIII in Patients With Severe Haemophilia A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GENA-21B
Record Dates: First submitted 2014-09-30; First posted 2014-10-06 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-12

CONDITIONS: Severe Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Human-cl rhFVIII (Experimental)
  Interventions: Biological: Human cl rhFVIII

INTERVENTIONS:
Biological: Human cl rhFVIII

SUMMARY:
The rationale of this study is to further fine-tune and individualize prophylactic treatment of patients with severe Haemophilia A with the goal of keeping the trough FVIII level above 1% between doses. Because trough FVIII levels are likely to be important predictors of the efficacy of prophylaxis, the focus of this study is on pharmacokinetic (PK) data.

ELIGIBILITY:
Inclusion Criteria:

* Severe Haemophilia A (FVIII:C < 1%)
* Male patients >= 18 years of age
* Previous treatment with a FVIII concentrate for at least 150 EDs
* Good documentation regarding dosing and bleeding frequency in the 6 months preceding study start
* Immunocompetence (CD4+ count > 200/uL)

Exclusion Criteria:

* Any coagulation disorder other than Haemophilia A
* Present of past FVIII inhibitor activity
* Severe liver or kidney disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig M Kessler, MD, Principal Investigator — Georgetown University
Locations (30):
- United States (9):
  - Octapharma Research Site, Sacramento, California
  - Octapharma Research Site, Aurora, Colorado
  - Octapharma Research Site, Washington D.C., District of Columbia
  - Octapharma Research Site, Miami, Florida
  - Octapharma Research Site, Chicago, Illinois
  - Octapharma Research Site, Indianapolis, Indiana
  - Octapharma Research Site, Memphis, Tennessee
  - Octapharma Research Site, Houston, Texas
  - Octapharma Research Site, Salt Lake City, Utah
- Canada (3):
  - Octapharma Research Site, Edmonton, Alberta
  - Octapharma Research Site, St. John's, Newfoundland and Labrador
  - McMaster University, Hamilton, Ontario
- University Hospital Centre Zagreb, Zagreb, Croatia
- Helsinki University Hospital, Helsinki, Finland
- France (5):
  - Centre Régional de Traitement de l'Hémophilie, Bron
  - CHU Estaing, Clermont-Ferrand
  - Centre Hospitalier Universitaire Félix Guyon, La Réunion
  - Centre Régional de Traitement de l'hémophilie, Nantes
  - Hôpital Purpan - Centre de Traitment Regional de l'Hemophilie Pole, Toulouse
- Japan (8):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Hospital of the Univ of Occupational and Environmental Health, Kitakyushu, Fukuoka
  - St. Marianna Univ School of Medicine Hospital, Kawasaki, Kanagawa
  - Nara Medical University Hospital, Kashihara, Nara
  - Gunma University Hospital, Maebashi
  - Osaka National Hospital, Osaka
  - Ogikubo Hospital, Tokyo
  - Teikyo University Hospital, Tokyo
- University Medical Center Groningen, Groningen, Netherlands
- PHI Institute of Transfusion Medicine of Republic of Macedonia, Skopje, North Macedonia
- University Medical Centre Ljubljana, Ljubljana, Slovenia

RESULTS

PARTICIPANT FLOW:
Groups:
- Human-cl rhFVIII: The study consisted of 3 phases:
  1. Pharmacokinetic (PK) Phase: 58 previously treated (≥150 exposure days) immunocompetent adults with severe hemophilia A without inhibitors patients started and completed the PK phase (PK population). Patients were treated with single dose of FVIII (60±5 IU/kg). One patient discontinued after single PK administration.
  2. Prophylactic Treatment Phase I: 57 patients started and 56 completed Phase I; Patients were treated prophylactically every other day or 3x/week with a dose of 30-40 IU/kg BW for 1-3 months until PK data had been analysed.
  3. Prophylactic Treatment Phase II: 56 patients started and 52 completed Phase II. Patients were treated prophylactically for 6 months using the dose and dosing interval based on individual PK data.
  All 58 patients were included in the safety (SAF) and the intention-to-treat (ITT) populations.
Period: Pharmacokinetic (PK) Evaluation Phase
Arm/Group | Human-cl rhFVIII
Started | 58
Completed | 58
Not Completed | 0
Period: Prophylactic Treatment Phase I
Arm/Group | Human-cl rhFVIII
Started | 57
Completed | 56
Not Completed | 1
Not completed — Lost to Follow-up | 1
Period: Prophylactic Treatment Phase II
Arm/Group | Human-cl rhFVIII
Started | 56
Completed | 52
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawn Consent | 1
Not completed — Did not attend completion visit | 1
Not completed — Discontinued medication | 1

BASELINE CHARACTERISTICS:
Groups:
- SAF/ITT Population: All patients who received at least one infusion of Human-cI rhFVIII
Arm/Group | SAF/ITT Population
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 39
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  Canada | 4
  Netherlands | 2
  United States | 23
  Japan | 11
  Finland | 4
  North Macedonia | 4
  Slovenia | 2
  France | 6
  Croatia | 2
Weight [Mean (Standard Deviation); unit: kg] | 77.0 (17.0)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.7 (5.0)
Hemophilia Joint Health Score [Mean (Standard Deviation); unit: units on a scale] — Joint health status will be assessed using the Hemophilia Joint Health Score (HJHS), which evaluates six index joints to produce a score between 0-124. Higher scores indicate worse joint health.
  units on a scale | 32.3 (20.2)
Blood group [Count of Participants; unit: Participants]
  O | 20
  A | 26
  AB | 1
  B | 7
  Unknown/missing | 4

OUTCOME MEASURES:

1. Primary Outcome: Annualized Total Bleeding Rate of Individually Tailored Prophylaxis
Description: Total annualized bleeding rate (ABR) of individually tailored prophylaxis (GENA-21b) compared to historical bleeding rate in patients having received on-demand treatment (GENA-01) with Human-cl rhFVIII
Time Frame: 6 months
Population: The analysis population comprised 56 patients who received at least one infusion of Human-cI rhFVIII for individualized prophylaxis in the GENA-21b trial. Their annualized bleeding rate was compared with those in patients from the completed GENA-01 trial who received only on-demand treatment.
Measure: Mean (Standard Deviation); unit: Bleeding events per year (ABR)
Groups:
- Individualized Prophylaxis in GENA-21b: Patients who received at least one infusion of Human-cI rhFVIII for individualized prophylaxis
- GENA-01: All patients receiving on-demand treatment with Human-cl rhFVIII in GENA-01
Arm/Group | Individualized Prophylaxis in GENA-21b | GENA-01
Number analyzed (Participants) | 56 | 22
Bleeding events per year (ABR) | 4.67 (6.46) | 58.08 (30.78)
Statistical Analysis 1: Comparison: Individualized Prophylaxis in GENA-21b vs GENA-01; Test type: Other — Confirmative one-sided one-sample Poisson-test; one-sided one-sample Poisson-test — A respective confirmative one-sided one-sample Poisson-test was used to demonstrate if the mean ABR in patients with individually tailored prophylaxis is at least 50% below the mean ABR rate in the GENA-01 trial; ABR = 4.87, 95% CI 2-sided [4.06 to 5.79] — A confidence interval of 97.5% for confirmative analysis was also used - the respective upper and lower limit CIs were 3.96-5.93
Statistical Analysis 2: Comparison: Individualized Prophylaxis in GENA-21b vs GENA-01; Test type: Other — Reduction of the annualized total bleeding rate (ABR) observed in the GENA-01 study vs. GENA-21B analyzed with a Negative Binomial regression model including a correction for overdispersion; p < 0.0001, Negative binomial regression model; Rate ratio = 11.89, 95% CI 2-sided [7.50 to 18.86]
Statistical Analysis 3: Comparison: Individualized Prophylaxis in GENA-21b vs GENA-01; Test type: Other — Reduction of the annualized total bleeding rate (ABR) observed in the GENA-01 study vs. GENA-21B analyzed with a Poisson regression model including a correction for overdispersion; p < 0.0001, Poisson regression model; Rate ratio = 10.14, 95% CI 2-sided [6.12 to 16.80]

2. Secondary Outcome: Annualized Spontaneous Bleeding Rate of Individually Tailored Prophylaxis
Description: Spontaneous annualized bleeding rate (ABR) of individually tailored prophylaxis (GENA-21b) compared to historical bleeding rate in patients having received on-demand treatment (GENA-01) with Human-cl rhFVIII
Time Frame: 6 months
Population: The analysis population comprised 56 patients who received at least one infusion of Human-cI rhFVIII for individualized prophylaxis in the GENA-21b trial. Their annualized spontaneous bleeding rate was compared with those in patients from the completed GENA-01 trial who received only on-demand treatment.
Measure: Mean (Standard Deviation); unit: Bleeding events per year (ABR)
Groups:
- Individualised Prophylaxis in GENA-21b: Patients who received at least one infusion of Human-cI rhFVIII for prophylaxis
Arm/Group | Individualised Prophylaxis in GENA-21b | GENA-01
Number analyzed (Participants) | 56 | 22
Bleeding events per year (ABR) | 2.98 (5.76) | 38.46 (28.07)
Statistical Analysis 1: Comparison: Individualised Prophylaxis in GENA-21b vs GENA-01; Test type: Other — A respective confirmative one-sided one-sample Poisson-test was used to demonstrate if the mean spontaneous ABR in patients with individually tailored prophylaxis is at least 50% below the mean ABR rate in the GENA-01 trial; One-sided one-sample Poisso; ABR = 3.12, 95% CI 2-sided [2.48 to 3.87]

3. Secondary Outcome: Annualized Total Bleeding Rate in Patients With 2x/Week (or Less) Prophylaxis
Description: Total annualized bleeding rate (ABR) in patients with 2x/week (or less) prophylaxis (GENA-21b) compared to historical bleeding rate in patients having received on-demand treatment (GENA-01) with Human-cl rhFVIII
Time Frame: 6 months
Population: The analysis population comprised 29 patients who received at least one infusion of Human-cI rhFVIII for individualized prophylaxis in the GENA-21b trial at intervals of 2x/week or less. Their annualized spontaneous bleeding rate was compared with those in patients from the completed GENA-01 trial who received only on-demand treatment.
Measure: Mean (Standard Deviation); unit: Bleeding events per year (ABR)
Groups:
- Prophylaxis 2x/Week or Less: Patients who received at least one infusion of Human-cI rhFVIII for prophylaxis and were treated with a prophylaxis infusion frequency of 2x/week or less
Arm/Group | Prophylaxis 2x/Week or Less | GENA-01
Number analyzed (Participants) | 29 | 22
Bleeding events per year (ABR) | 4.82 (6.98) | 58.08 (30.78)
Statistical Analysis 1: Comparison: Prophylaxis 2x/Week or Less vs GENA-01; Test type: Other — A respective confirmative one-sided one-sample Poisson-test was used to demonstrate if the mean ABR in patients with 2x/week prophylaxis or less with individually tailored prophylaxis is at least 50% below the mean ABR rate in the GENA-01 trial; One-sided one-sample Poisson-test; ABR = 5.03, 95% CI 2-sided [3.90 to 6.39] — A confidence interval of 97.5% for confirmative analysis was also used - the respective upper and lower limit CIs were 3.76-6.60

4. Secondary Outcome: Median Prophylactic Dosing Interval
Description: Median over median actual dosing intervals between two prophylactic treatments per patient. The median time (hours) between two prophylactic doses of Human-cl rhFVIII in the prophylactic treatment Phase II per patient
Time Frame: 6 months
Population: The analysis population comprised 56 patients who received at least one infusion of Human-cI rhFVIII for individualized prophylaxis in the GENA-21b trial.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Prophylaxis: Patients who received at least one infusion of Human-cI rhFVIII for prophylaxis
Arm/Group | Prophylaxis
Number analyzed (Participants) | 56
hours | 83.9 [53.5 to 96.1]

5. Secondary Outcome: Mean Prophylactic Dosing Interval
Description: Mean over mean actual dosing intervals between two prophylactic treatments per patient. The mean time (hours) between two prophylactic doses of Human-cl rhFVIII in the prophylactic treatment Phase II per patient
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prophylaxis
Number analyzed (Participants) | 56
hours | 83.0 (22.37)

6. Secondary Outcome: AUC Divided by the Dose (AUCnorm) of Human-cl rhFVIII
Description: AUCnorm of Human-cl rhFVIII measured using the one-stage (OS) assay
Time Frame: Before injection (within 1 h before injection) and up to 72 h (± 2 h) after the end of injection
Population: The PK-PP population contained all patients in the PK analysis population who completed the initial PK sampling phase of the trial without significantly violating the inclusion/exclusion criteria or other aspects of the protocol considered to potentially affect the PK results.
Measure: Mean (Standard Deviation); unit: hr*IU/mL/(IU/kg)
Groups:
- PK Evaluation: PK-PP population
Arm/Group | PK Evaluation
Number analyzed (Participants) | 47
hr*IU/mL/(IU/kg) | 0.302 (0.116)

7. Secondary Outcome: In-vivo Recovery (IVR) of Human-cl rhFVIII
Description: IVR of Human-cl rhFVIII measured using the one-stage (OS) assay and will be determined from the FVIII level before the infusion and the peak level after the infusion of Human-cl rhFVIII
Time Frame: Before injection (within 1 h before injection) and up to 72 h (± 2 h) after the end of injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: % per IU/kg
Arm/Group | PK Evaluation
Number analyzed (Participants) | 47
% per IU/kg | 1.775 (0.421)

8. Secondary Outcome: Half Life (t1/2) of Human-cl rhFVIII
Description: T1/2 of Human-cl rhFVIII measured using the one-stage (OS) assay
Time Frame: Before injection (within 1 h before injection) and up to 72 h (± 2 h) after the end of injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PK Evaluation
Number analyzed (Participants) | 47
hours | 15.725 (4.029)

9. Secondary Outcome: Mean Residence Time (MRT) of Human-cl rhFVIII
Description: MRT of Human-cl rhFVIII measured using the one-stage (OS) assay
Time Frame: Before injection (within 1 h before injection) and up to 72 h (± 2 h) after the end of injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PK Evaluation
Number analyzed (Participants) | 47
hours | 20.762 (5.997)

10. Secondary Outcome: Clearance (CL) of Human-cl rhFVIII
Description: CL of Human-cl rhFVIII measured using the one-stage (OS) assay
Time Frame: Before injection (within 1 h before injection) and up to 72 h (± 2 h) after the end of injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/hr/kg
Arm/Group | PK Evaluation
Number analyzed (Participants) | 47
mL/hr/kg | 3.859 (1.670)

11. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Human-cl rhFVIII
Description: Vss of Human-cl rhFVIII measured using the one-stage (OS) assay
Time Frame: Before injection (within 1 h before injection) and up to 72 h (± 2 h) after the end of injection
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | PK Evaluation
Number analyzed (Participants) | 47
mL/kg | 72.901 (16.454)

12. Secondary Outcome: Usage of Human-cl rhFVIII (FVIII IU/kg BW Per Week Per Patient)
Description: Average weekly consumption of Human-cl rhFVIII reported as IU/kg BW per week per patient was determined during individualized prophylactic treatment
Time Frame: 6 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: IU/kg per week
Groups:
- Prophylaxis: Patients who received at least one infusion of Human-cI rhFVIII for prophylaxis in Phase III
Arm/Group | Prophylaxis
Number analyzed (Participants) | 56
IU/kg per week | 83.7 (25.7)

13. Secondary Outcome: Number of Patients With Adverse Events (AEs)
Description: AEs were documented at each (scheduled or unscheduled) study visit. Severity and seriousness of all AEs were documented by the investigator according to pre-defined criteria
Time Frame: At each study visit over the study duration (7-9 months)
Population: The SAF population included 58 patients who received at least one infusion of Human-c1 rhFVIII in the GENA-21b trial
Measure: Count of Participants; unit: Participants
Arm/Group | SAF/ITT Population
Number analyzed (Participants) | 58
Participants
  AE | 34
  No AE | 24

ADVERSE EVENTS:
Time Frame: At each study visit over the study duration (7-9 months)
Arm/Group | SAF/ITT Population
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 4/58
Other Adverse Events (participants affected / at risk) | 34/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAF/ITT Population (N=58)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Subdural haematoma (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SAF/ITT Population (N=58)
Nasopharyngitis (Infections and infestations) | 12
Influenza (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Diarrhea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pyrexia (General disorders) | 4
Headache (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Octapharma agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Octapharma supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial. Octapharma also reserves the right to review data prior to publishing and provide comments/changes within a certain time period.

DOCUMENTS (2):
  • Study Protocol (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02256917/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02256917/SAP_003.pdf